CLINICAL TRIAL: NCT01897077
Title: The Safety and Efficacy of a Peanut Immunotherapy Dissolving Film for Peanut Allergy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study product manufacturing suspended due to manufacturing problems, before initiation of study intervention.
Sponsor: Johns Hopkins University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00042409
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Peanut Allergy
Keywords: Food Allergy; Peanut; Sublingual Immunotherapy
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peanut Allergic (Experimental): Only one intervention will be given. Peanut allergic study subjects, will receive gradually increasing doses of the dissolving peanut film.
  Interventions: Drug: Peanut Dissolving Film
- Healthy Volunteers (Active Comparator): Healthy volunteers will receive active peanut dissolving films in an expedited manner in order to determine safety dissolving films.
  Interventions: Drug: Peanut Dissolving Film

INTERVENTIONS:
Drug: Peanut Dissolving Film

SUMMARY:
The purpose of this study is to determine if a new method of administration of peanut sublingual immunotherapy, a dissolving peanut film, is effective.

DETAILED DESCRIPTION:
Peanut allergy is a common problem with no current treatment. Recent studies have shown some success with oral or sublingual immunotherapy for the treatment of food allergy. Oral treatment, which requires very high doses, is associated with a small but appreciable risk of systemic reactions. Sublingual immunotherapy, which utilizes much smaller doses, is safer but constraints inherent in the available methods of sublingual administration have limited the utility of this method. Typically sublingual immunotherapy for food allergy has used either fresh foods or a simple liquid extract. These methods are not optimized for practicality or dwell duration in the mouth, and, thus far, dosing has been limited by the ability to make concentrated extracts and by the volume of extract that can be applied to the sublingual space. This study is being conducted to determine if a dissolving peanut extract film, will improve efficacy for immunotherapy for peanut allergy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years
* Provide signed informed consent
* Using appropriate birth control if subject is female and of child bearing age
* Are available for the study duration

Healthy Volunteers Only

* Regularly consume a meal sized portion (5 grams) of peanut at least twice per month during the proceeding 6 months

Peanut Allergic Subjects Only

* Have a history of symptomatic reactivity to peanut
* Have a positive skin prick test
* Have a positive oral food challenge to peanut at a cumulative dose of less than 1 grams of peanut protein
* Have self-injectable epinephrine available at home

Exclusion Criteria:

* Have a history of severe anaphylaxis to peanut, defined as hypoxia, hypotension or neurological compromise as a result of ingestion of peanut.
* Have a history of intubation related to asthma
* Are pregnant or lactating
* Have a viral Upper Respiratory Infection (URI) or gastroenteritis within 7 days of Oral food challenge
* Have pulmonary function tests <80% of predicted (FEV1) or clinical history consistent with more than moderate persistent asthma
* Are currently taking greater than medium dose inhaled corticosteroid (>500 mcg/day fluticasone or fluticasone equivalent)
* Are unable to discontinue antihistamines for 5 days for long acting and 3 days for short acting prior to skin testing or food challenges
* Have used systemic corticosteroids within 4 weeks prior to baseline visit
* Are receiving omalizumab, beta-blocker, Angiotensin Converting Enzyme (ACE) inhibitor or tricyclic antidepressant therapy. Subjects need to be off omalizumab for 6 months.
* Have history of oral cancer.
* Use oral tobacco (i.e., chew tobacco)
* Have a chronic disease (other than asthma, atopic dermatitis or rhinitis) requiring therapy (e.g., heart disease, diabetes)
* Have participated in any interventional study for treatment of a food allergy in the past 12 months
* Have a history of eosinophilic esophagitis
* Have a severe reaction at initial double blind placebo-controlled food challenge, defined as either:

  * Life-threatening anaphylaxis, or
  * Reaction requiring hospitalization

Healthy Volunteers Only

* History of any allergy to peanut

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2013-02-03 (Actual); Study Completion 2013-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, MD, Principal Investigator — Johns Hopkins University; Corinne Keet, MD, MS, Principal Investigator — Johns Hopkins University; Hugh Sampson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mount Sinai School of Medicine, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Peanut Allergic: Only one intervention will be given. Peanut allergic study subjects, will receive gradually increasing doses of the dissolving peanut film.
  Peanut Dissolving Film.
  No subjects were enrolled before termination.
- Healthy Volunteers: Healthy volunteers will receive active peanut dissolving films in an expedited manner in order to determine safety dissolving films.
  Peanut Dissolving Film
  5 subjects received the active film.
Period: Overall Study
Arm/Group | Peanut Allergic | Healthy Volunteers
Started | 0 | 5
Completed | 0 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study ended prematurely before any peanut allergic subjects were enrolled.
Groups:
- Peanut Allergic: Only one intervention will be given. Peanut allergic study subjects, will receive gradually increasing doses of the dissolving peanut film.
  Peanut Dissolving Film
- Healthy Volunteers: Healthy volunteers will receive active peanut dissolving films in an expedited manner in order to determine safety dissolving films.
  Peanut Dissolving Film
- Total: Total of all reporting groups
Arm/Group | Peanut Allergic | Healthy Volunteers | Total
Number analyzed (Participants) | 0 | 5 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 5 | 5
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 3 | 3
  Male |  | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 2 | 2
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 2 | 2
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects That Discontinue the Study for Treatment Related Reasons
Description: No healthy volunteers discontinued the study for treatment related reasons. No active participants enrolled.
Time Frame: 18 months
Population: There were no peanut allergic subjects enrolled because the study ended prematurely due to manufacturing issues with the study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Allergic | Healthy Volunteers
Number analyzed (Participants) | 0 | 5
Participants |  | 0

2. Secondary Outcome: The Proportion of Subjects Who Are Able to Tolerate the Full 10 Gram Peanut Protein Challenge at the Completion of the Study
Description: For peanut allergic subjects only
Time Frame: 18 months
Population: No participants were analyzed for this secondary outcome because data was not collected due to early termination of the study
Arm/Group | Peanut Allergic | Healthy Volunteers
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Effects With Therapy
Time Frame: 18 months
Population: No participants were analyzed for this secondary outcome in the peanut allergic group because data was not collected due to early termination of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Allergic | Healthy Volunteers
Number analyzed (Participants) | 0 | 5
Participants | 0 | 0

4. Secondary Outcome: The Rate of Medication Use With Therapy
Description: For peanut allergic subjects only.
Time Frame: 18 months
Population: No participants were analyzed for this secondary outcome because no data for the outcome was collected due to early termination of the study
Arm/Group | Peanut Allergic | Healthy Volunteers
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Changes in Biomarkers (Peanut Specific Immunoglobulin E (IgE) and Immunoglobulin G (IgG), Basophil Reactivity, and Salivary Biomarkers) From Baseline to the End of Therapy
Description: Only in peanut allergic subjects
Time Frame: 18 months
Population: as for outcome 2
Arm/Group | Peanut Allergic | Healthy Volunteers
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Serious Adverse Events With Dosing
Time Frame: 18 months
Population: No participants were analyzed for this secondary outcome in the peanut allergic group because no data was collected due to early termination of the study
Measure: Number; unit: participants
Arm/Group | Peanut Allergic | Healthy Volunteers
Number analyzed (Participants) | 0 | 5
participants |  | 0

ADVERSE EVENTS:
Time Frame: 1 month for healthy volunteers
Description: Because the study ended prematurely, no peanut allergic subjects were enrolled, so there were no subjects at risk for serious adverse events, all-cause mortality or other adverse events.
Arm/Group | Peanut Allergic | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/5
Other Adverse Events (participants affected / at risk) | 0/0 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes